

### Statistical Analysis Plan

24 Feb 2021

# Title of trial: A Multi-Center, Randomized, Assessor-Blind, Controlled Trial Comparing the Occurrence of Major Adverse Cardiovascular Events (MACEs) in Patients with Prostate Cancer and Cardiovascular Disease Receiving Degarelix (GnRH Receptor Antagonist) or Leuprolide (GnRH Receptor Agonist) NCT number: NCT02663908 Sponsor trial code: 000108 Date:

Date: 24 Feb 2021 E-Statistical Analysis Plan-19595; Ver.7.0 Supersedes: 6.0 

### STATISTICAL ANALYSIS PLAN

A Multi-Center, Randomized, Assessor-Blind, Controlled Trial Comparing the Occurrence of Major Adverse Cardiovascular Events (MACEs) in Patients with Prostate Cancer and Cardiovascular Disease Receiving Degarelix (GnRH antagonist) or Leuprolide (LHRH agonist)

### 000108

**IND Number:** 051222

Investigational Medicinal Product: Degarelix powder and solvent for solution for injection

Leuprolide acetate 22.5 mg 3 month depot

**Indication:** Prostate cancer

Phase: 3b

**Date of issue:** 24 February 2021

Version: 7.0

The information in this document is confidential and is proprietary to Ferring Pharmaceuticals A/S or another company within the Ferring Group. It is understood that information in this document shall not be disclosed to any third party, in any form, without prior written consent of an authorised officer of Ferring Pharmaceuticals A/S or another company within the Ferring Group

**Authors:** 

# **Change log**

| Version<br>No. | Effective<br>Date | Reason for the Change / Revision Supersedes | |
|---|---|---|---|
| 1 | Dec 16 – 2015 | Original SAP | Not Applicable |
| 2 | Dec 18 – 2015 | Format Change only. No content was changed. | |
| 3 | | The list of major protocol deviations in Section 5 was updated to reflect the changes to the clinical trial protocol introduced with clinical trial protocol amendment #01. | Version 2.0 |
| 4 | Mar 28 - 2017 | To update the SAP in order to relect the revised eligibility criteria for the trial based on recommendations from the Steering Committee and changes made to the trial protocol in agreement with the US Food and Drug Administration (FDA) following review of the Clinical Trial Protocol Amendment number 01, dated 21 September 2016. | |
| 5 | Nov-18-2019 | The list of key secondary endpoints has been revised, and sensitivity endpoint "Time from randomization to the first confirmed (adjudicated) occurrence of cardiovascular death, non-fatal myocardial infarction or non-fatal stroke" has been added to the list, and the testing strategy has been changed from Holm's to a fixed. Also, PP analyses have been reduced to primary and exploratory endpoints. | Version 4.0 "Time from med iovascular retion or nonnel list, and mged from yses have |

| 6 | Sep 30 - 2020 | Due to the trial being terminated early, the SAP was updated. The following changes has been made to the SAP: | Version 5.0 |
|---|---|---|---|
| | | - Due to site errors in randomizations, the FAS will be used instead of ITT in order to present "correct" denominator in tables. | |
| | | - Planned interim analyses have been cancelled. | |
| | | - Various changes to analyses no longer affected by the expected interim. | |
| | | - Sensitivity analyses of the primary endpoint including PP analyses have been cancelled. | |
| | | - Some analyses have been reduced (not removed) as deemed unnecessarily extensive, others have been slightly altered. | |
| | | - Analyses regarding markedly abnormal laboratory values have been cancelled as deem unnecessary by pharmacovigilance. | |
| 7 | Feb-24-2021 | Sensitivity analyses added to primary analysis. Slight rewording of some endpoints. Endpoint "Total number of emergency room (ER) visit events over the duration of the trial" changed to "Total number of CV-related emergency room (ER) visit events over the duration of the trial". Treatment switch definition updated | |
| | | according to data collected. Important deviations to be summarized. General rewordings and clarifications added. | |


# Signed Agreement on Statistical Analysis Plan

| Author: Statistician, Global Biometrics |
|---|
| The statistical analysis plan was reviewed by, |
| Urology, Global Clinical Development, Ferring Pharmaceuticals A/S |
| Urology, Global Clinical Development, Ferring Pharmaceuticals A/S |
| Statistician, Global Biometrics, Ferring Pharmaceuticals A/S |
| Statistical Programmer, Global Biometrics, Ferring Pharmaceuticals A/S |
| Clinical Trial Manager, Global Clinical Operations, Ferring Pharmaceuticals A/S |
| Pharmacovigilance physician, Global Pharmacovigilance, Ferring Pharmaceuticals A/S |
| Medical Writer, Global Medical Writing, Ferring Pharmaceuticals A/S |
| The statistical analysis plan was reviewed and approved (signed electronically) by, |
| Global Biometrics, Ferring Pharmaceuticals A/S |

### TABLE OF CONTENTS

| 1 | <b>Intr</b><br>1.1 | oduction | |
|---|---|---|---|
| 2 | Tria | l Objectives and Endpoints | |
| _ | 2.1 | Objectives | |
| | | 2.1.1 Primary Objective | |
| | | 2.1.2 Secondary Objectives | 10 |
| | | 2.1.3 Exploratory Objectives | 11 |
| | 2.2 | Endpoints | 11 |
| | | 2.2.1 Primary Endpoint | 11 |
| | | 2.2.2 Secondary Endpoints | 11 |
| | | 2.2.3 Exploratory Endpoints | 12 |
| 3 | | l design | 13 |
| | The | following section details the original trial design. However, the trial was terminated due to feasibility problems, with only 545 patients randomized and 14 of those with positively | |
| | | adjudicated events. Hence, many of these sections no longer apply | 13 |
| | 3.1 | General Design Considerations | |
| | 3.1 | Determination of Sample Size. | |
| | 3.2 | 3.2.1 Fixed Trial Design. | |
| | | 3.2.2 Adjustments for Futility Analyses | |
| | | 3.2.3 Adjustments for Sample Size Re-Estimation | |
| 4 | Pati | ent Disposition | |
| 5 | | cool Deviations | |
| 6 | | lysis Sets | |
| U | 6.1 | Intention-To-Treat Analysis Set | |
| | 6.2 | Full Analysis Set. | |
| | 6.3 | Safety Analysis Set | |
| _ | | | |
| 7 | | l Population | |
| | 7.1 | Demographics and Other Baseline Characteristics | |
| | | 7.1.1 Demographics | |
| | | 7.1.2 Vital Signs at Baseline | |
| | | 7.1.3 History and Stage of Prostate Cancer | |
| | | 7.1.5 Laboratory Efficacy / Pharmacodynamic Parameters at Baseline | 20 |
| | 7.2 | Laboratory Efficacy / I harmacodynamic I arameters at Baseniie | 20<br>■ 20 |
| | 7.2 | 7.2.1 | 20 |
| | 7.3 | | 20 |
| | 7.4 Physical Examination | | |
| 8 | Exp | osure and Treatment Compliance | 22 |
| | 8.1 | Extent of Exposure. | |
| | 8.2 | Treatment Compliance | 22 |
| 9 | Effic | cacy | 23 |
| | 9.1 | General Considerations | 23 |


| | 9.2 | Primary | Endpoint | | 24 |
|---|---|---|---|---|---|
| | | 9.2.1 | Primary E | ndpoint Analysis | 24 |
| | | 9.2.2 | Sensitivity | Analyses | 25 |
| | | | 9.2.2.1 | Sensitivity Analysis: Time from randomization to the first confirmed (adjudicated) occurrence of non-fatal myocardial infarction, non-fatal stroke, non-fatal unstable angina requiring hospitalization, or all-cause death | 25 |
| | | | 9.2.2.2 | Sensitivity Analysis: Time to first confirmed occurrence of a MACE related adverse event (MI SMQ (broad); Central nervous system hemorrhages and cerebrovascular conditions SMQ (broad); all-cause death) | 25 |
| | | | 9.2.2.3 | Sensitivity Analysis: Total occurrence of (adjudicated) myocardial infarction, stroke, and all-cause death | 25 |
| | | | 9.2.2.4 | Sensitivity Analysis pertaining to treatment discontinuation or initiation of prohibited therapies related to hormonal therapy | |
| | 9.3 | Seconda | ry Endpoint | S | |
| | | 9.3.1 | | n randomization to the first confirmed (adjudicated) occurrence of cular-related death, non-fatal myocardial infarction or non-fatal stroke | 26 |
| | | 9.3.2 | | n Randomization to the first (adjudicated) occurrence of the individual ats of the MACE composite endpoint | 27 |
| | | 9.3.3 | | n randomization to the first confirmed (adjudicated) unstable angina hospitalization | 28 |
| | | 9.3.4 | | n Randomization to Death Due to Any Cause | 28 |
| | | 9.3.5 | | n Randomization to confirmed (adjudicated) Cardiovascular-Related | 28 |
| | | 9.3.6 | Time from | n Randomization to Failure in Progression-Free Survival | 29 |
| | | 9.3.7 | | ne levels at day 28, 168 and 336 in patients treated with degarelix and | 30 |
| | | 9.3.8 | | ber of Cardiovascular-Related Hospitalizations over the duration of the | 30 |
| | | 9.3.9 | | ber of Coronary Artery By-Pass Grafting or Percutaneous Coronary on Procedures over the duration of the trial | 30 |
| | | 9.3.10 | | ber of Cardiovascular-Related Emergency Room Visit Events over the duration of the trial | 31 |
| | | 9.3.11 | | e in Quality Adjusted Life Year (QALY) During One Year of Treatment | |
| | | 9.3.12 | _ | om Baseline in Mean Total and QoL International Prostate Symptom ing One Year of Treatment | 32 |
| | | 9.3.13 | | om Baseline in the Mean Duke Activity Status Index and Cardiac Questionnaire Score during One Year of Treatment | 32 |
| | 9.4 | Explora | | nts | |
| | | 9.4.1 | | n First Adjudicated MACE to Second Confirmed Adjudicated MACE | |
| | | 9.4.2 | | | 34 |
| | | 9.4.3 | | | _ |
| | | | | | 34 |
| 10 | | • | | | |
| | 10.1 | General | Considerati | ons | 35 |


| 10. | .2 Adverse | | | |
|---|---|---|---|---|
| | 10.2.1 | | Treatment-Emergent Adverse Events | |
| | 10.2.2 | | Adverse Events | |
| 10. | 10.3 Safety Laboratory Variables | | | |
| | 10.3.1 Summary Statistics | | | |
| | 10.3.2 Laboratory Variable Changes Relative to Normal Range | | | |
| | 10.3.3 | _ | S | |
| 4.0 | 10.3.4 | • | | |
| 10. | , | , | | |
| | 10.4.1 | _ | | |
| | | | Summary Statistics | |
| | | | Markedly Abnormal Changes | |
| | | | Data Listings | |
| 11 Int | terim Analy | sis | | 40 |
| 12 De | viations fro | m Protocol A | nalysis | 41 |
| 14 Ta | bles, Listin | gs and Figure | S | 43 |
| Appen | | | bnormal Vital Signs and Electrocardiograms (ECGs) | |
| | | · | | |
| Appendix 2 SMQs for AE Medical History of Special Interest | | | | |
| | | | and MedDRA terms for disease progression | 46 |
| Appen | dix 4 | ATC codes | and MedDRA terms for Prohibited Therapy | |
| Appen<br>Appen | | ATC codes | and MedDRA terms for Prohibited Therapylar Endpoint Definitions | |
| | | ATC codes | | |
| Appen | | ATC codes Cardiovascu | | |
| Appen | dix 5<br>OF TABL | ATC codes Cardiovascu | ılar Endpoint Definitions | |
| Append | dix 5 OF TABLE Sampl | ATC codes Cardiovascu | tions (Number of Events Rounded Upwards) | |
| Appendus LIST (Table 1 | OF TABLE Sample Marke | ATC codes Cardiovasco ES e Size Calcula dly abnormal | tions (Number of Events Rounded Upwards) | |
| Appendum LIST (Table 1 Table 2 | OF TABL<br>Sampl<br>Marke<br>Abnor | ATC codes Cardiovasco ES e Size Calcula dly abnormal control of the codes of the | tions (Number of Events Rounded Upwards) | |
| Appendix LIST (Table 1 Table 2 Table 3 | OF TABLE Sample Market Abnor | ATC codes Cardiovascu ES e Size Calcula dly abnormal mal Criteria for | tions (Number of Events Rounded Upwards) | |
| Appendix LIST (Table 1 Table 2 Table 3 Table 4 | OF TABLE Sample Market Abnor Cardio | ATC codes and Cardiovascular Eventes Events | tions (Number of Events Rounded Upwards) | |
| Appendicular Appen | OF TABLE Sample Market Abnor Cardio Diabet ATC O | ES e Size Calcula dly abnormal mal Criteria fo vascular Even es Events | tions (Number of Events Rounded Upwards). 15 Criteria for Vital Signs* 44 or Quantitative ECG Data. 44 tts. 45 androgens 46 | |
| Appendicular Appen | OF TABLE Sample Market Abnor Cardio Diabet ATC O | ES e Size Calcula dly abnormal mal Criteria fo vascular Even es Events Codes for Anti odes for Addi | tions (Number of Events Rounded Upwards) | |
| Appendent LIST (Table 1 Table 2 Table 3 Table 4 Table 5 Table 6 Table 7 | OF TABLE Sample Market Abnor Cardio Diabet ATC O MedD | ES e Size Calcula dly abnormal mal Criteria fo vascular Even es Events Codes for Anti odes for Addi RA Codes (pr | tions (Number of Events Rounded Upwards) | |
| Appendix App | OF TABL Sampl Market Abnor Cardio Diabet ATC O MedD MedD MedD | ES e Size Calcula dly abnormal mal Criteria fo vascular Even es Events Codes for Anti odes for Addi RA Codes (pr RA Codes (pr RA Codes (pr | tions (Number of Events Rounded Upwards) | |
| Appendent LIST (Table 1 Table 2 Table 3 Table 4 Table 5 Table 6 Table 7 Table 8 Table 9 Table 1 | OF TABLE Sample Market Abnor Cardio Diabet ATC O MedD MedD Of dise | ES e Size Calcula dly abnormal mal Criteria fo vascular Even es Events Codes for Anti odes for Addi RA Codes (pr RA Codes (pr RA Codes (pr esase progression | tions (Number of Events Rounded Upwards) | |
| Appendent LIST (Table 1 Table 2 Table 3 Table 5 Table 6 Table 7 Table 8 Table 9 Table 1 Table 1 | OF TABLE Sample Market Abnor Cardio Diabet ATC of MedD MedD of dise 1 ATC of | ES e Size Calcular dly abnormal emal Criteria for vascular Events Codes for Antiodes for Addi RA Codes (pro RA Codes (pro) | tions (Number of Events Rounded Upwards) | |
| Appendent LIST (Table 1 Table 2 Table 3 Table 4 Table 5 Table 6 Table 7 Table 8 Table 9 Table 1 | OF TABLE Sample Market Abnor Cardio Diabet ATC of MedD MedD of dise 1 ATC of | ES e Size Calcular dly abnormal emal Criteria for vascular Events Codes for Antiodes for Addi RA Codes (pro RA Codes (pro) | tions (Number of Events Rounded Upwards) | |
| Appendent LIST (Table 1 Table 2 Table 3 Table 4 Table 5 Table 6 Table 7 Table 8 Table 9 Table 1 Table 1 Table 1 | OF TABLE Sample Market Abnor Cardio Diabet ATC of MedD MedD of dise 1 ATC of | ES e Size Calcula dly abnormal mal Criteria fo vascular Even es Events Codes for Anti odes for Addi RA Codes (pr RA Codes (pr RA Codes (pr esse progression odes for prohi RA code (pref | tions (Number of Events Rounded Upwards) | |


### 1 Introduction

This document describes the planned statistical analyses for Trial 000108.

### 1.1 Abbreviations

ADT Androgen Deprivation Therapy
AIC Akaike Information Criterion
ANCOVA Analysis of Covariance

ATC Anatomical Therapeutic Chemical

AUC Area Under the Curve BMI Body Mass Index

CABG Coronary Artery by-pass Grafting
CAQ Cardiac Anxiety Questionnaire
CDF Cumulative Distribution Function
CEC Clinical Events Classification

CI Confidence Interval CV Cardiovascular

CVD Cardiovascular Disease
DASI Duke Activity Status Index

DSMB Data and Safety Monitoring Board

ECG Electrocardiogram

EQ-5D-5L EuroQol Group 5 Dimensions Questionnaire

ER Emergency Room FAS Full Analysis Set FPR False Positive Rate

GnRH Gonadotropin-Releasing Hormone

HbA<sub>1c</sub> Hemoglobin A<sub>1c</sub>

HRQL Health-Related Quality of Life

IMP Investigational Medicinal Product

IPCW Inverse Probability of Censoring Weights IPSS International Prostate Symptom Score

ITT Intention-to-Treat

KMMI Kaplan-Meier Multiple Imputation

LHRH Luteinizing Hormone Releasing Hormone

LUTS Lower Urinary Tract Symptoms
MACE Major Adverse Cardiovascular Event

MedDRA Medical Dictionary for Regulatory Activities

MRI Magnetic Resonance Imaging

PCA Prostate cancer

PCI Percutaneous Coronary Intervention

PFS Progression-Free Survival

PP Per Protocol

PRO Patient Reported Outcome PSA Prostate-specific Antigen

PT Preferred Term

QALY Quality Adjusted Life Year

Date: 24 Feb 2021 E-Statistical Analysis Plan-19595; Ver.7.0 Supersedes: 6.0


ROC Receiver Operating Characteristics

SOC System Organ Class
TPR True Positive Rate

WHO World Health Organization
WLW Wei – Lin – Weissfeld


### 2 Trial Objectives and Endpoints

### 2.1 Objectives

### 2.1.1 Primary Objective

• The primary objective is to assess the effect of a GnRH receptor antagonist (degarelix) on the risk of occurrence of MACEs (a composite of death due to any cause, non-fatal myocardial infarction or non-fatal stroke) as compared to a GnRH receptor agonist (leuprolide) in patients with prostate cancer and concomitant CVD

### 2.1.2 Secondary Objectives

### CV and Death Related Objectives

- To assess the rate of specific MACEs (individual components of the composite MACE endpoint), i.e. myocardial infarction (fatal, non-fatal), stroke (fatal, non-fatal), in patients randomized to degarelix versus leuprolide
- To assess the rate of unstable angina requiring hospitalization (fatal, non-fatal), in patients randomized to degarelix versus leuprolide
- To assess the risk of death due to any cause in patients randomized to degarelix versus leuprolide
- To assess the rate of cardiovascular (CV)-related death in patients randomized to degarelix versus leuprolide

### **Prostate Cancer-Related Objectives**

- To monitor testosterone levels at Day 28, 168 and 336 in the degarelix and leuprolide treatment groups
- To evaluate the progression-free survival (PFS) failure rates (defined as either death, radiographic disease progression<sup>a</sup>, introduction of additional therapy related to prostate cancer<sup>b</sup> or prostate-specific antigen [PSA] failure<sup>c</sup>, whichever is first) in the degarelix and leuprolide treatment groups
  - a. One or more new metastatic skeletal lesions observed on bone scan; one or more new metastatic extraskeletal lesions at least 1.5 cm in greatest dimension visible on computed tomography or magnetic resonance imaging (MRI) scan as confirmed by the Investigator.
  - b. Additional therapy includes radiation, anti-androgens (except for initial symptomatic flare protection) and second-line treatment.
  - c. PSA failure is defined as an increase in serum PSA of 50%, and at least 5 ng/mL, compared to nadir, measured on two consecutive occasions at least 2 weeks a part.
- To compare the effects of degarelix with leuprolide with regards to local urinary tract and prostate cancer-related symptoms with the International Prostate Symptom Score (IPSS) questionnaire

### Health Economics and Patient Reported Outcome (PRO) Objectives

• To compare the effects of degarelix with leuprolide with regards to healthcare resource use

Date: 24 Feb 2021 E-Statistical Analysis Plan-19595; Ver.7.0 Supersedes: 6.0 

- To compare the effects of degarelix with leuprolide with regards to health status through the EuroQol Group 5 Dimensions Questionnaire (EQ-5D-5L)
- To compare the effects of degarelix with leuprolide with regards to functional capacity and Quality of Life (QoL) through the Duke Activity Status Index (DASI)
- To compare the effects of degarelix with leuprolide with regards to heart-focused anxiety through the Cardiac Anxiety Questionnaire (CAQ)

### Safety Objective

• To evaluate and compare the overall safety and tolerability of degarelix with leuprolide

### 2.1.3 Exploratory Objectives

• To compare the effects of degarelix with leuprolide with regards to a second confirmed (adjudicated) occurrence of the composite MACE endpoint, in the subgroup of patients that survived the first CV event



### 2.2 Endpoints

### 2.2.1 Primary Endpoint

• Time from randomization to the first confirmed (adjudicated) occurrence of the composite MACE endpoint

### 2.2.2 Secondary Endpoints

### Key Secondary Endpoints

- Time from randomization to the first confirmed (adjudicated) occurrence of CV-related death, non-fatal myocardial infarction or non-fatal stroke
- Time from randomization to confirmed (adjudicated) CV-related death
- Time from randomization to the first confirmed (adjudicated) myocardial infarction

### Other CV and Death-Related Endpoints

- Time from randomization to the first confirmed (adjudicated) stroke
- Time from randomization to the first confirmed (adjudicated) unstable angina requiring hospitalization
- Time from randomization to death due to any cause

### Prostate Cancer-related Endpoints


- Testosterone levels at Days 28, 168 and 336 in the degarelix and leuprolide treatment groups
- Time from randomization to failure in PFS
- Changes from baseline in IPSS Total and Qol scores

### Health Economics and Patient-Reported Outcomes Endpoints

- Total number of CV-related hospitalization events over the duration of the trial
- Total number of coronary artery by-pass grafting (CABG) or percutaneous coronary intervention (PCI) procedures over the duration of the trial
- Total number of CV-related emergency room (ER) visit events over the duration of the trial
- Change in utility, based on EQ-5D-5L
- Changes from baseline in DASI Global score
- Changes from baseline in CAQ Global score and score per domain

### Safety Endpoints

- Incidence and intensity of adverse events
- Changes in vital signs

### 2.2.3 Exploratory Endpoints

first CV event

occurrence of the composite MACE endpoint in the subgroup of patients that survived the

Time from first adjudicated non-fatal MACE to a second confirmed (adjudicated)


### 3 Trial design

The following section details the original trial design. However, the trial was terminated due to feasibility problems, with only 545 patients randomized and 14 of those with positively adjudicated events. Hence, many of these sections no longer apply.

### 3.1 General Design Considerations

This is a multi-center, randomized, assessor-blind, controlled trial to compare MACEs in patients with prostate cancer and concurrent CVD receiving either monthly treatment with degarelix or leuprolide 3-month depot for 1 year. Patients will be screened within 8 to 21 days prior to randomization for compliance with the inclusion and exclusion criteria. A trial design diagram is provided in Figure 1.



Figure 1 Trial Design Diagram

Patients will be randomized to one of the two treatments in a 1:1 ratio stratified by age group (<75 and ≥75 years of age) and region (North America, other). After randomization, the management of prostate cancer is intended to reflect standard-of-care. Monitoring for possible MACEs will occur throughout the trial applying a specific Clinical Events Classification (CEC) process ensuring blinding of the event assessors.

### 3.2 Determination of Sample Size

The primary objective is to assess the effect of degarelix on the risk of MACEs (a composite of death due to any cause, non-fatal myocardial infarction or non-fatal stroke) occurring during a 1-year period as compared to treatment with leuprolide in patients with prostate cancer and concomitant CVD.

The observed one-year event rates for primary MACE endpoint are 5.3% and 12.1% for degarelix and LHRH agonist, respectively, in the global patient population with prior CVD were derived from a post-hoc analysis of degarelix safety data. This would correspond to an unadjusted treatment-

Date: 24 Feb 2021 E-Statistical Analysis Plan-19595; Ver.7.0 Supersedes: 6.0 

related hazard ratio of 0.42. (In comparison, the adjusted hazard ratio is 0.39 (95% confidence interval [CI] = [0.21; 0.71]).) Furthermore, based upon the re-assessment of the potential CV events captured in the degarelix safety data by an independent cardiologist, the one-year event probability for CV event or death due to any cause are 4.8% and 9.3% for degarelix and leuprolide respectively. This corresponds to an unadjusted hazard ratio of 0.50 (in comparison, the adjusted hazard ratio is 0.48 (95% confidence interval is [0.23,0.87]). Accounting for the uncertainty in the post-hoc analysis of the global pooled data and the re-assessment of the potential CV events by a single independent cardiologist, the one-year event rates for sample size calculations are set to 5.1% and 10.2% for degarelix and leuprolide, respectively. This corresponds to a hypothesized hazard ratio of 0.49.

### 3.2.1 Fixed Trial Design

Given the alternative hypothesis, a power of 80% and a signficiance level of 5%, the expected number of events required at the final analysis is 61. The sample size required for achieving this number of events assumes that all patients are followed-up for primary outcome (MACEs) for 12 months (28 days each) after start of treatment and an annual drop-out rate of 5%. Assuming these characteristics a total sample size of 811 patients is required.

### 3.2.2 Adjustments for Futility Analyses

One interim analysis is planned after 50% of the confirmed, adjudicated MACE endpoints have been collected. One of the objectives of the interim analysis is to test whether there is any reason to stop early for futility. The futility bound expressed in terms of the hazard ratio is 0.78. That is, if the observed hazard ratio is >0.78 the Data and Safety Monitoring Board (DSMB) may suggest to stop the trial due to futility. The futility bounds are non-binding. Due to the possibility to stop early for futility the power is deflated (risk of stopping a successful trial is inflated), and to reinstall the power at 80% the number of required events is inflated to 66 and the total number of patients to 876.

The trial will not be stopped early due to an overwhelming treatment benefit, but in order to implement the trial design, an alpha-spending function will be used with nearly zero spending of alpha at the interim analysis,  $\alpha < 0.0001$  (e.g. trial will not be stopped early for efficacy).

### 3.2.3 Adjustments for Sample Size Re-Estimation

The conditional power for different sample size increases will be evaluated at the interims using SAS. In case of a sample size increase, the final test statistic is adjusted by using the normal inverse method in order to protect the two-sided Type I error rate at 5%.

The sample size calculations are performed with ADDPLAN™ 6, licensed by ADDPLAN, Inc., an Aptiv Solutions company and presented in Table 1.


Table 1 Sample Size Calculations (Number of Events Rounded Upwards)

| Information<br>Rate | Stop for futili | ty/No eviden | ce reject H <sub>0</sub> | Successful trial (Reject H <sub>0)</sub> | g gnant | Power | Events |
|---|---|---|---|---|---|---|---|
| | Test Statistic | Hazard<br>Ratio | Conditional<br>Power | Test Statistic | α spent | | |
| 50% | ≤ 0.7 | ≥0.78 | ≤8.5% | - | < 0.0001 | - | 33 |
| 100% | ≤1.96 | ≥ 0.61 | - | ≥ 1.96 | 0.025 | 80% | 66 |

- Assuming constant hazards,  $\lambda_{degarelix} = 0.0523/year$   $\lambda_{leuprolide} = 0.1076/year$
- 5% drop out rate in each arm
- 1:1 randomization ratio

When d, the number of events, has been observed, the approximate relationship between the standardized test statistic, Z, and the hazard ratio (HR) as given in (Jennison and Turnbull, 2000) is,

$$Z \approx log(HR^{-1})\sqrt{d/4}$$

For reasons of interpretation, both Z and the hazard ratio are reported in design tables.

Date: 24 Feb 2021 E-Statistical Analysis Plan-19595; Ver.7.0 Supersedes: 6.0 

### 4 Patient Disposition

All patients screened and randomized will be accounted for. All post-randomization discontinuations will be summarized by time of, and reason for, discontinuation. The number of patients screened and not randomized will be presented with the reason(s) for screen failure.

Special attention should be paid to those patients who discontinue treatment with investigational medicinal product (IMP) and start an alternative treatment during the trial, including the dates corresponding to going off the randomized drug, i.e. the date of the last injection and the start of a new treatment, i.e. the date the new treatment was initiated.

In addition, the breakdown of the overall disposition of patients by age group (<75 years of age, ≥75 years of age) and region following the design (stratification) of the trial will be provided. Also, the number of patients screened and randomized, overall and by age group (<75 years of age, ≥75 years of age) and region will be provided.

1- Kaplan–Meier (1-KM) plots of the time to early discontinuation, as well as the time to treatment discontinuation or initiation of prohibited therapies related to hormonal therapy, will be displayed per treatment arm. In addition, time to early discontinuation by reason for discontinuation and treatment arm will be presented by cumulative incidence function curves. Differences in discontinuation rates and treatment discontinuation or initiation of prohibited therapies related to hormonal therapy rates between treatment groups will be tested using the Log Rank test ( $\alpha$ =0.05, two-sided).

Date: 24 Feb 2021 E-Statistical Analysis Plan-19595; Ver.7.0 Supersedes: 6.0


### 5 Protocol Deviations

As no PP analyses are planned, there will be no classification of 'minor'/'major' events, reflecting potential impact on efficacy endpoints due to protocol violations.

In order to reflect general (i.e. not specifically related to impact on efficacy) protocol adherence important deviations will be summarized by treatment group and category, and listed by subject for the Full Analysis Set.


### 6 Analysis Sets

### **6.1** Intention-To-Treat Analysis Set

The Intention-to-Treat (ITT) analysis set consists of all randomized patients, and will be analysed based on the planned (randomized) treatment.

### 6.2 Full Analysis Set

The Full Analysis Set (FAS) consists of all randomized and treated patients (who received at least one dose of IMP), and will be analysed based on the planned (randomized) treatment.

### 6.3 Safety Analysis Set

The Safety analysis set consists of all treated patients (who received at least one dose of IMP), and will be analysed based on the actual treatment received.


### 7 Trial Population

All tables will be presented for the FAS.

### 7.1 Demographics and Other Baseline Characteristics

Categorical data will be summarized using numbers and percentages. The percentages are based on the total number of patients with a corresponding assessment. Continuous data will be presented, for example, using the number of patients (N), mean and standard deviation, median, minimum and maximum. All baseline characteristics will be listed.

### 7.1.1 Demographics

### 7.1.2 Vital Signs at Baseline

### 7.1.3 History and Stage of Prostate Cancer

A summary table of history and stage of PCA will be presented, containing the following information:

- Gleason score (as defined below)
- Stage of prostate cancer (TNM classifications, as defined below)
- ECOG performance score

The following pathological stages will be recorded and summarized by treatment group, age (<75 years and  $\ge 75$  years) and region:

The Gleason score is calculated as the sum of the Gleason grade of the primary and secondary patterns. The following categories will be presented:

- 2-4
- 5-6
- 7-10

The stage of prostate cancer, based on the TNM classification, includes the following categories:

• Localised: T½ & (NX or N0) & M0,

• Locally Advanced: [T<sup>3</sup>/<sub>4</sub> & (NX or N0) & M0], or [N1 & M0],

• Metastatic: M1

| • | Not classifiable: | Results from T, N, and M categories that could not be resolved to Localised, Locally Advanced, or Metastatic |
|---|---|---|
| 1.5 | | cy / Pharmacodynamic Parameters at Baseline |
| seli | ne variables will be s | ummarized by treatment, age (<75 years and ≥75 years) and region. |

Date: 24 Feb 2021 E-Statistical Analysis Plan-19595; Ver.7.0 Supersedes: 6.0


### 7.4 Physical Examination

Patients with abnormalities at any screening, baseline, or post-baseline visit will be listed with all physical examination evaluations.


### 8 Exposure and Treatment Compliance

All tables will be presented for the FAS.

### 8.1 Extent of Exposure

The cumulated dose administered to each patient will be determined and summarized descriptively. For patients discontinuing the trial early, are lost to follow-up or initiate treatment with an ADT other than Degarelix or Leuprolide, their cumulated dose will be calculated up until the time of early discontinuation/lost to follow-up/treatment iniation.

### 8.2 Treatment Compliance

Treatment compliance will be presented from data listings. Patients not receiving the scheduled dose will be listed by center, sorted by treatment group and patient number.


### 9 Efficacy

The following sections detail the planned analyses in the protocol. Any changes to the planned analysis in the protocol are described in Section 12.

### 9.1 General Considerations

The analysis of efficacy will be performed for the FAS (unless otherwise specified). For the purpose of this CV outcome study, patients prematurely discontinuing from treatment will be followed-up for the occurrence of MACE events based on monthly telephone interviews. Unless otherwise stated, time to event endpoints will be censored at the time of treatment discontinuation, initiation of prohibited therapies related to hormonal therapy, lost to follow-up/withdrawal from the study or day 336, whichever occurs first. Initiation of prohibited therapy related to hormonal therapy includes the following:

- Surgical castration or other hormonal manipulation in addition to the IMPs
- Anti-androgens for combined androgen blockade (anti-androgen use for initial flare protection is allowed for a maximum period of up to 28 days after randomization)
- Estrogens
- Megestrol acetate
- Ketoconazole
- Abiraterone
- Enzalutamide
- Any additional hormonal therapy initiated as a combination therapy with the IMP

The associated ATC and MedDRA codes for the above prohibited therapies are provided in Table 11 and Table 12. Hypothesis tests will be two-sided at a significance level of 5% and missing data will not be imputed. 95% confidence limits and the associated p-values will be presented for estimates of the treatment effect comparing degarelix to leuprolide for all regression analyses.

| For the purposes of | this trial, | |
|---------------------|-------------|---|
| _ | | |
| | | • |



### 9.2 Primary Endpoint

### 9.2.1 Primary Endpoint Analysis

The primary endpoint, the time from randomization to the first adjudicated occurrence of the composite MACE endpoint in the two treatment groups, will be analyzed using the Kaplan-Meier estimator of the survival function and the log-rank test, stratified for age (<75 and ≥75 years of age) and region and based on the FAS.

Pseudo SAS code for Kaplan-Meier/log-rank test:

```
PROC LIFETEST DATA=<DATA> PLOTS=SURVIVAL();

TIME AVAL*CNSR(1);

STRATA <STRAT1 STRAT2> /GROUP=ARMN TEST=LOGRANK;
RUN;
```

The hazard ratio, comparing the hazard rate of the distribution of the time from randomization to the MACE composite endpoint between the degarelix and leuprolide arms, will be estimated based on the stratified Cox regression model, stratified by age-group and region and including treatment as a factor. The variance estimate of the log hazard ratio will be obtained from the inverse of the observed information matrix for the partial likelihood. An approximate 95% CI for the hazard ratio will be calculated by exponentiation of the 95% CI for the log hazard ratio. Although, the score test for this stratified Cox Regression model is equivalent to the stratified log-rank test, (Kalbfleisch and Prentice, 2002), the (Wald based) 95% CI may not be fully consistent with the stratfied log-rank test. The latter, however, defines the success of the trial. More precisely, the trial will be declared positive if a statistically significant (at two-sided 5% significance level) reduction in the hazard rate of the time from randomization to the composite MACE endpoint is demonstrated in the FAS based on the stratified log-rank test, for patients randomized to degarelix compared to leuprolide.

TLF Figure: Primary Endpoint: Time to First Adjudicated MACE – FAS


### 9.2.2 Sensitivity Analyses

# 9.2.2.1 Sensitivity Analysis: Time from randomization to the first confirmed (adjudicated) occurrence of non-fatal myocardial infarction, non-fatal stroke, non-fatal unstable angina requiring hospitalization, or all-cause death

Time from randomization to the first confirmed (adjudicated) occurrence of non-fatal myocardial infarction, non-fatal stroke, non-fatal unstable angina requiring hospitalization, or all-cause death is defined similarly as the primary endpoint with the addition of cardiovascular events unstable angina requiring hospitalization. Also, the endpoint will be analyzed as for the primary endpoint.

# 9.2.2.2 Sensitivity Analysis: Time to first confirmed occurrence of a MACE related adverse event (MI SMQ (broad); Central nervous system hemorrhages and cerebrovascular conditions SMQ (broad); all-cause death)

Time to first confirmed occurrence of a MACE related adverse event is defined as for the primary endpoint with events being; any adverse event within the broad SMQ term 'myocardial infarction', any adverse event within broad SMQ term 'Central nervous system hemorrhages and cerebrovascular conditions' or all-cause death. Also, the endpoint will be analyzed as for the primary endpoint.

# 9.2.2.3 Sensitivity Analysis: Total occurrence of (adjudicated) myocardial infarction, stroke, and all-cause death

Total occurrence of myocardial infarction (MI), stroke and all-cause death is defined as the total number of events (MI, stroke or death) occurring over the duration of the trial.

The endpoint will be compared between treatment groups using a negative binomial model. The estimated treatment difference with a 95% confidence interval will be presented.

# 9.2.2.4 Sensitivity Analysis pertaining to treatment discontinuation or initiation of prohibited therapies related to hormonal therapy

For the purposes of this sensitivity analysis, patients will NOT be censored at the time of treatment discontinuation or initiation of prohibited therapies related to hormonal therapy. Rather, information pertaining to all observed occurrences of the first adjudicated MACE event in patients randomized in the study will be used. Patients will be censored at lost to follow-up/withdrawal from study or day 336, whichever occurs first.

### 9.3 Secondary Endpoints

If the primary analysis is significant at the two-sided Type I error-level of 5% the testing of the secondary endpoints will proceed as described below.

### Key Secondary Analyses

The following analyses are included in the family of key secondary analyses:

Date: 24 Feb 2021 E-Statistical Analysis Plan-19595; Ver.7.0 Supersedes: 6.0 

- Time from randomization to the first confirmed (adjudicated) occurrence of CV-related death, non-fatal myocardial infarction or non-fatal stroke
- Time from randomization to confirmed (adjudicated) CV-related death
- Time from randomization to the first confirmed (adjudicated) myocardial infarction

The key secondary endpoints will be controlled for multiplicity (to ensure the family wise error rate is protected at a two-sided 5% Type I error-level) using a fixed-sequence testing method. The order of the testing sequence is as follows:

- 1. Time from randomization to the first confirmed (adjudicated) occurrence of CV-related death, non-fatal myocardial infarction or non-fatal stroke
- 2. Time from randomization to confirmed (adjudicated) CV-related death
- 3. Time from randomization to the first confirmed (adjudicated) myocardial infarction

The remaining secondary endpoints will be analyzed without controlling for multiplicity.

### Other Secondary Analyses

- Time from randomization to the first confirmed (adjudicated) stroke
- Time from randomization to first confirmed (adjudicated) unstable angina requiring hospitalization
- Time from randomization to death due to any cause
- Time from randomization to failure in PFS
- Testosterone levels at Days 28, 168 and 336 in the degarelix and leuprolide treatment groups
- Total number of CV-related hospitalizations over the duration of the trial
- Total number of CABG or PCI procedures over the duration of the trial
- Total number of CV-related ER visit events over the duration of the trial
- Changes from baseline in Health-Related Quality of Life (HRQL) as measured by EQ-5D-5L, during the course of treatment period
- The difference in QALY during one year of treatment with degarelix compared to leuprolide
- The change from baseline in the mean DASI and CAQ score during one year of treatment with degarelix compared to leuprolide
- The change from baseline in the mean total and QoL IPSS score during oneyear of treatment with degarelix compared to leuprolide

# 9.3.1 Time from randomization to the first confirmed (adjudicated) occurrence of cardiovascular-related death, non-fatal myocardial infarction or non-fatal stroke

This endpoint is identical to the primary endpoint, only counting CV-related deaths, and not all cause deaths as failures. The time measured in days, from randomization to first confirmed (adjudicated) occurrence of CV-related death, non-fatal myocardial infarction or non-fatal stroke,

will be analyzed using the Kaplan-Meier estimator of the survival function and the log-rank test of the null hypothesis of equal hazard functions, stratified by age group and region. The p-value of the two-sided log-rank test with significance level of 5% will be presented along with plots of the estimated survival functions for the two treatment groups, stratified by age group and region. The treatment effect of degarelix will be further examined by fitting a stratified Cox regression model. The model will include treatment as a factor, be adjusted for the baseline CV risk factors as appropriate and stratified by age-group and region. The 95% confidence limits and associated p-value for the hazard ratio comparing treatment with degarelix to leuprolide will be presented.

TLF Table: Secondary Endpoint: CV Death + MI + Stroke - FAS

TLF Figure: Secondary Endpoint: CV Death + MI + Stroke - FAS

# 9.3.2 Time From Randomization to the first (adjudicated) occurrence of the individual components of the MACE composite endpoint

Time from randomization to the first adjudicated occurrence of the individual components of the MACE composite endpoint is defined as the number of days from randomization to the first adjudicated myocardial infarction/stroke. The occurrence of the components of the MACE composite endpoint will be adjudicated by the external independent CEC Committee. In order to correctly assess the treatment effect associated with degarelix with respect to the time to individual components of the MACE composite endpoint, it is necessary to account for the competing risk, death due to other causes. The above components of the MACE composite endpoint will be analyzed separately. The log-rank test stratified by age-group and region will be used to examine the null hypothesis of equal cumulative cause specific hazard functions. The p-value of the two-sided log rank test with significance level of 5% will be presented along with the plots of the estimated cumulative cause specific hazard functions for both treatments obtained from the Nelson-Aalen estimator, stratified by age group and region.

TLF Table: Secondary Endpoint: Time to First Adjudicated Myocardial Infarction - FAS

TLF Figure: Cumulative Cause Specific Hazard Function for Time to First Adjudicated Myocardial Infarction – FAS

TLF Table: Secondary Endpoint: Time to First Adjudicated Stroke - FAS

TLF Figure: Cumulative Cause Specific Hazard Function for Time to First Adjudicated Stroke – FAS


# 9.3.3 Time from randomization to the first confirmed (adjudicated) unstable angina requiring hospitalization

Time from randomization to the first adjudicated occurrence of unstable angina requiring hospitalization will be analyzed in the same manner as the individual components of the MACE primary endpoint, specified in Section 9.3.2.

TLF Table: Secondary Endpoint: Time to First Adjudicated Unstable Angina Requiring Hospitalization – FAS

TLF Figure: Cumulative Cause Specific Hazard Function for Time to First Adjudicated Unstable Angina Requiring Hospitalization – FAS

### 9.3.4 Time From Randomization to Death Due to Any Cause

Time from randomization to death due to any cause (overall survival, OS), is defined as the number of days from randomization to death. The time measured in days, from randomization to death due to any cause, will be analyzed using the Kaplan-Meier estimator of the survival function and the log-rank test of the null hypothesis of equal hazard functions, stratified by age group and region. The p-value of the two-sided log-rank test with significance level of 5% will be presented along with plots of the estimated survival functions for the two treatment groups, stratified by age group and region. The treatment effect of degarelix will be further examined by fitting a stratified Cox regression model for the time to death from any cause. The model will include treatment as a factor, be adjusted for the baseline CV risk factors as appropriate and stratified by age-group and region. The 95% confidence limits and associated p-value for the hazard ratio comparing treatment with degarelix to leuprolide will be presented.

TLF Table: Secondary Endpoint: Time to Death Due to Any Cause – FAS

TLF Figure: Survivor Function for Time to Death Due to Any Cause – FAS

### 9.3.5 Time from Randomization to confirmed (adjudicated) Cardiovascular-Related Death

Time from randomization to adjudicated CV-related death, is defined as the number of days from randomization to the date of the adjudicated CV-related death. The cause of death will be adjudicated by the external independent CEC Committee. Undetermined deaths will be presumed and analyzed as non-cardiovascular deaths. In order to correctly assess the treatment effect associated with degarelix with respect to the time to CV-related death, it is necessary to account for the competing risk, death due to other causes. The time measured in days, from randomization to the adjudicated CV-related death, will be analyzed using the Nelson-Aalen estimator of the cumulative cause specific hazard function and the log rank test of the null hypothesis of equal cumulative cause specific hazard functions, stratified by age group and region. The p-value of the two-sided log rank test with significance level of 5% will be presented along with plots of the cumulative cause specific hazard functions for the two treatment groups, stratified by age group and region. The treatment effect of degarelix will be further examined by fitting a stratified Cox-type


regression model for the cause specific hazard function associated with CV-related death. The model will include treatment as a factor, be adjusted for the baseline CV risk factors as appropriate and stratified by age-group and region. The 95% confidence limits and associated p-value for the cause specific hazard ratio comparing treatment with degarelix to leuprolide will be presented.

TLF Table: Secondary Endpoint: Time to Adjudicated Cardiovascular-related Death - FAS

TLF Figure: Cumulative Cause Specific Hazard Function for Time to Adjudicated Cardiovascular-related Death – FAS

### 9.3.6 Time from Randomization to Failure in Progression-Free Survival

Progression-free survival (PFS) is a composite endpoint consisting of the following conditions:

- Death
- Radiographic disease progression defined as one or more new metastatic skeletal lesions observed on bone scan; one or more new metastatic extra-skeletal lesions at least 1.5 cm in greatest dimension visible on computed tomography or magnetic resonance imaging scan as confirmed by the Investigator.
- Introduction of additional therapy related to prostate cancer treatment including radiation, anti-androgens and second-line treatment. (ATC and MedDRA codes for disease progression are included in Appendix 3)
- PSA failure defined as the time from randomization to the second occasion (must be at least two weeks apart from the first and correspond to consecutive measurements) in which the PSA value fulfills the following criteria:
  - I. An absolute increase of  $\geq 5$  ng/ml above nadir and
  - II. An increase of > 50 % of nadir

Time to PFS failure is therefore defined as the time, measured in days, from randomization to the first occurrence of one of the above composite endpoint criteria. Patients discontinuing from treatment/withdrawn from the study will be censored at the time of discontinuation/withdrawal. Time to PFS failure will be analyzed using the Kaplan-Meier estimator of the survival function, the Cox regression model for the hazard rate and the log-rank test of the null hypothesis of equal hazard functions, stratified by age group and region. The p-value of the two-sided stratified log-rank test with significance level of 5% will be presented along with plots of the estimated survival functions for the two treatment groups, stratified by age group and region. The estimated hazard ratio and the associated 95% confidence interval and p-value comparing the treatment with Degarelix to Leuprolide will also be presented.

TLF Table: Secondary Endpoint: Time to PFS Failure - FAS

TLF Figure: Survivor Function for Time to PFS Failure - FAS


# 9.3.7 Testosterone levels at day 28, 168 and 336 in patients treated with degarelix and leuprolide

The proportion of patients castrated at day 28, 168 and 336 will be presented by treatment group, along with the number of patients with testosterone measurements at each assessment. Castration is defined as testosterone levels  $\leq 0.5$  ng/mL. Further, the proportion of patients castrated at both day 28 and 168, as well as at all three visits will be presented along with the number of patients with assessments at each of the corresponding times. For patients discontinuing treatment during the trial, any testosterone data collected after the date of discontinuation will be excluded from the analysis.

# TLF Table: Secondary Endpoint: Probability of testosterone levels remaining at castrate levels – FAS

### 9.3.8 Total number of Cardiovascular-Related Hospitalizations over the duration of the trial

The total number of CV-related hospitalizations over the duration of the trial is defined as the number of hospitalizations due to CV-related adverse events, observed during the 12 month follow-up period for each patient.

The number of CV-related hospitalizations will be analyzed using a negative binomial model. The dependent variable will be the number of CV-related hospitalizations. The model will include a factor variable for treatment, the baseline count of CV-related hospitalizations (if available) as a covariate and will be further adjusted by including the logarithm of the number of days of follow-up for each patient as an offset. The inclusion of the offset term systematically adjusts the estimate of the treatment effect for potential differences in the duration of follow-up between patients. The model will further be adjusted for age-group and region. The estimated treatment difference with a 95% confidence interval will be presented.

# TLF Table: Secondary Endpoint: Number of CV-related hospitalizations over the duration of the trial – FAS

# 9.3.9 Total number of Coronary Artery By-Pass Grafting or Percutaneous Coronary Intervention Procedures over the duration of the trial

The total number of CABG or PCI procedures observed over the duration of the trial will be analyzed in the same manner as the total number of CV-related hospitalizations, outlined in Section 9.3.8.

TLF Table: Secondary Endpoint: Number of CABG or PCI over the duration of the trial – FAS


# 9.3.10 Total number of Cardiovascular-Related Emergency Room Visit Events Observed over the duration of the trial

The total number of CV-related ER visit events observed over the duration of the trial for each patient will be analyzed in the same manner as the total number of CV-related hospitalizations, outlined in Section 9.3.8.

TLF Table: Secondary Endpoint: Number of Cardiovascular-related emergency room visits over the duration of the trial – FAS

### 9.3.11 Difference in Quality Adjusted Life Year (QALY) During One Year of Treatment

The EQ-5D-5L questionnaire can be used to estimate the QALY. The QALY is a measure of the value of health outcomes. Since health is a function of length of life and QoL, the QALY was developed as an attempt to combine the value of these attributes into a single index number. The basic idea underlying the QALY is simple: it assumes that a year of life lived in perfect health is worth 1 QALY (1 Year of Life × 1 Utility value = 1 QALY) and that a year of life lived in a state of less than this perfect health is worth less than 1. The QALY is derived as a cumulative measure for the treatment duration as the AUC of the time versus the index value. The AUC will be calculated using the trapezoidal rule for each of the visits values in relation to the baseline.

A detailed derivation of the QALY:

- The EQ-5D-5L health state is converted into a single index value. The index values are country specific and we will use the value sets for the USA (http://www.euroqol.org/home.html.).
- 2) The QALY at the end of the trial is derived as the cumulative AUC for the index value as a function of time during the 12 months of treatment. This will be calculated as:

$$AUC = \sum_{i=1}^{i} \left( \frac{index_{(i-1)} + index_i}{2} \right) \times Time_{(i-(i-1))}$$

Where i=1, 2 and 3 for the corresponding visits at month 6, 11 and 12. The value, i=0, corresponds to baseline.

Time is measured as the actual number of days from baseline date of EQ-5D to each of the post-baseline EQ-5D Questionnaire completion dates during the 12 month trial.

The QALY at Visit 13 will be calculated for any patients who have a non-missing baseline index value. That is, any patients who are missing the EQ5D index value at baseline will not have a QALY measurement. Last observation carried forward principle will be used for missing measurements at Visit 8 or Visit 13 using only post-baseline values. The EQ5D index value will be carried forward to the planned visit date in order to calculate the QALY at 12 months. For patients with missing index value at Visit 8, but with known index value either at Visit 13 or 14, the QALY will be calculated as the AUC from baseline up to the next known visit.

The mean QALY at the end of the trial (12 months [1 month=28 days]) will be summarized by treatment arm and compared using an analysis of covariance (ANCOVA) model, where the QALY is the dependent variable and adjusted for treatment, age-group and region respectively.

# 9.3.12 Change from Baseline in Mean Total and QoL International Prostate Symptom Score during One Year of Treatment

The severity of lower urinary tract symptoms (LUTS) will be investigated using the total IPSS score. IPSS is a questionnaire containing eight questions regarding incomplete emptying, frequency, intermittency, urgency, weak stream, straining and nocturia and one question relating to the quality of life. Each question is assigned a total score on a scale from 0 to 5. The total IPSS score is then calculated as the summation over the responses for question 1 to 7.

The eighth question regarding QoL is in relation to urinary symptoms denoted IPSS-QoL. The response to this question is analyzed separately and not included in the IPSS total score.

Missing values will not be imputed for this endpoint. If responses are missing to one or more of questions 1-7, the IPSS total score is considered missing as well. Results will be presented based on the observed cases.

Changes from baseline in the IPSS total score and QoL score will be compared between treatments longitudinally using repeated measures analysis of covariance (ANCOVA) with the change from baseline as the dependent variable and the baseline score as a covariate, treatment, age-group, region and visit as factors, including treatment by visit interaction term, assuming the working correlation matrix has the unstructured form implemented in SAS PROC MIXED. Based on the repeated measures ANCOVA model, the two-sided 95% confidence limits of the adjusted treatment contrasts and associated p-values will be provided.

### TLF Table: Secondary Endpoint: IPSS - FAS

# 9.3.13 Change from Baseline in the Mean Duke Activity Status Index and Cardiac Anxiety Questionnaire Score during One Year of Treatment

The DASI and CAQ will be assessed at baseline (Visit 2), Visit 8, 14 and at the End-of-Trial visit. The change from baseline in DASI total score as well as CAQ total and domain scores will be compared between treatments longitudinally using repeated measures ANCOVA with the change from baseline as the dependent variable and the baseline score as a covariate, treatment, age-group, region and visit as factors, including treatment by visit interaction term, assuming the working correlation matrix has the unstructured form implemented in SAS PROC MIXED. Based on the ANCOVA model, the two-sided 95% confidence limits of the adjusted treatment contrasts and associated p-values will be provided.

TLF Table: Secondary Endpoint: The change in the mean DASI Score during one-year of treatment-FAS


# TLF Table: Secondary Endpoint: The change from baseline in the mean CAQ Score during one-year of treatment – FAS

### 9.4 Exploratory Endpoints

### 9.4.1 Time from First Adjudicated MACE to Second Confirmed Adjudicated MACE

The exploratory efficacy endpoint, time from the first adjudicated MACE to a second confirmed (adjudicated) occurrence of the composite MACE endpoint, is aimed at further investigating the risk of CVD outcomes among prostate cancer patients treated with degarelix or LHRH agonist.

Only patients who have experienced one non-fatal MACE, will be considered at risk for a second MACE. The event time of interest will be the number of days from the first adjudicated non-fatal MACE until the second MACE. The endpoint will be analyzed via a Cox-type proportional intensity model. In essence the analysis is akin to the proposed conditional analysis of (Prentice, 1981) with a modification made based on the definition of the composite MACE endpoint. The model will include treatment as a factor, be a swell as stratified by age-group and region. Based on the Cox-type proportional intensity model, the two-sided 95% confidence limit of the adjusted relative rate for the treatment effect of degarelix compared to leuprolide will be provided alongside the associated p-value. Significant results will be interpreted cautiously, as randomization will not provide protection against imbalances between the two groups in potential confounders that are not explicitly adjusted for in the model. The treatment effect of degarelix compared to leuprolide with respect to the rate of MACEs will be further explored via an Andersen-Gill model (Andersen and Gill, 1982). The risk set for the Andersen-Gill model includes all patients who are under

observation and at-risk for a MACE, i.e. the Andersen-Gill model incorporates information from all

Pseudo SAS code for implementing Andersen-Gill model

PROC PHREG DATA=<DATA> COVS(AGGREGATE);

MODEL (TSTART, TSTOP)\*CNSR(1) = ARMN;

ID=USBJID;

RUN;

Note, in the above SAS code for the Andersen-Gill model, the robust standard errors are calculated by including the COVS(AGGREGATE) statement in the first line. Alternatively, model based standard errors could be returned by replacing the COVS(AGGREGATE) option with COVM.

TLF Table: Exploratory Endpoint: Time From First Non-Fatal adjudicated MACE to a Second Confirmed Occurrence of a MACE – FAS

observed MACEs.

Date: 24 Feb 2021 E-Statistical Analysis Plan-19595; Ver.7.0 Supersedes: 6.0 

### 10 Safety

### 10.1 General Considerations

Safety parameters will be evaluated for the safety dataset.

### 10.2 Adverse Events

Adverse events will be coded using MedDRA version 17.1 or later.

For adverse events, missing values will be treated as missing, except for causality, intensity, seriousness, and outcome of adverse events. A worst-case approach will be used: if causality is missing, the adverse event will be regarded as related to the IMP; if the intensity of an adverse event is missing, the adverse event will be regarded as severe; if seriousness is missing, the adverse event will be regarded as serious; if onset date is missing, it will be assumed to be the first day of dosing; if outcome is missing, and no date of outcome is present, the outcome is regarded as 'Not Recovered'.

An adverse event with the causal relationship to IMP judged as 'No reasonable possibility' is categorized as unrelated to IMP. An adverse event with the causal relationship to IMP judged as a 'reasonable possibility' is categorized as related to IMP and as an adverse drug reaction.

Treatment-emergent adverse events will be presented in summary tables and listings. The definition of a treatment-emergent adverse event is provided in Section 10.2.1.

### 10.2.1 Overview of Treatment-Emergent Adverse Events

Adverse events will be regarded as 'pre-treatment' if they occur between screening and the initial injections with IMP. Adverse events which occur in the time interval from initial dosing to 3 months after (1 month=28 days) last dosing of IMP will be considered to be 'treatment-emergent'. Adverse events will be regarded as 'post-treatment' if they occur 3 months (1 month=28 days) or more after the last dosing of IMP.

An adverse event overview summary table will be prepared including the number of patients reporting an adverse event, the percentage of patients (%) with an adverse event, and the number of events (E) reported, for the following categories:

- Treatment-emergent adverse events
- Deaths
- Serious adverse events
- Adverse events leading to withdrawal
- Severe and life threatening adverse events
- Adverse drug reactions

TLF Table: Overall summary of treatment-emergent adverse events – Safety
#### 10.2.2 Incidence of Adverse Events

Treatment-emergent adverse events will be summarized in a table by MedDRA SOC and Preferred Term (PT). The Table will display the total number of patients reporting an adverse event, the percentage of patients (%) with an adverse event, and the number of events (E) reported. Adverse events will be presented by SOC sorted alphabetically and PT sorted in decreasing frequency of occurrence.

For each treatment the following counts are done:

- For number of patients experiencing a particular event, counting will be done by patient and not by event. This is valid for both SOC and PT, i.e., a patient will only be counted once in each SOC and once within each PT.
- For total number of events, counting will be done by event. This is valid for both SOC and PT, i.e., an event occurring more than once for the same patient will be counted for each occurrence.

Summary tables will be prepared for:

- All adverse events
- Adverse events with an incidence  $[\geq 5\%]$  of patients in any treatment group
- Adverse events by causality (related/unrelated)
- Adverse events leading to death
- Adverse events by intensity
- Serious adverse events
- Adverse events leading to withdrawal

Supporting data listings will be provided for:

- All adverse events sorted by center and patient no.
- All adverse events sorted by MedDRA PT
- Serious adverse events
- Adverse events leading to death
- Adverse events leading to withdrawal.

In addition, tables summarizing all the treatment-emergent adverse events by MedDRA SOC and PT displaying the total number of patients reporting an adverse event, the percentage of patients (%) with an adverse event, and the number of events (E) reported will be provided.

TLF Table: Incidence of all adverse events by MedDRA System Organ Class and Preferred Term – Safety Analysis Set

TLF Table: Incidence of treatment-emergent non-serious adverse events (>5% cut-off) by MedDRA System Organ Class and Preferred Term – Safety Analysis Set

TLF Table: Incidence of all adverse events by causality, MedDRA System Organ Class and Preferred Term – Safety Analysis Set

TLF Table: Incidence of adverse events leading to death by MedDRA System Organ Class and Preferred Term – Safety Analysis Set

TLF Table: Incidence of all adverse events by intensity, MedDRA System Organ Class and Preferred Term – Safety Analysis Set

TLF Table: Incidence of serious adverse events by MedDRA System Organ Class and Preferred Term – Safety Analysis Set

TLF Table: Incidence of adverse events leading to withdrawal by MedDRA System Organ Class and Preferred Term – Safety Analysis Set

TLF Table: Incidence of treatment-emergent adverse events by MedDRA System Organ Class and Preferred Term – Safety Analysis Set

TLF Table: Incidence of treatment-emergent adverse drug reactions by MedDRA System Organ Class and Preferred Term - Safety Analysis Set

TLF Table: Incidence of treatment-emergent adverse events leading to discontinuations by MedDRA System Organ Class and Preferred Term - Safety Analysis Set

TLF Table: Incidence of treatment-emergent serious adverse events by MedDRA System Organ Class and Preferred Term – Safety Analysis Set

TLF Listing: Listings of all adverse events sorted by center and patient no.

TLF Listing: Listings of all adverse events sorted by MedDRA Preferred Term

TLF Listing: Listings of all serious adverse events

TLF Listing: Listings of all adverse events leading to death

TLF Listing: Listings of all adverse events leading to withdrawal

## 10.3 Safety Laboratory Variables

Baseline for all laboratory analyses will be the values obtained at the last assessment prior to the first dose of the IMP. Treatment-emergent laboratory data will include tests completed after the first dose of IMP through the residual time of drug effect. End of trial will include the last post-baseline observation during the trial.

## 10.3.1 Summary Statistics

Mean change and mean percentage (%) change from baseline to the end of trial will be presented for each laboratory variable. In addition, descriptive statistics, i.e., the number of patients with data,


mean (standard deviation), median, minimum, and maximum values, will be presented for observed values and change from baseline at each time-point for each laboratory variable.

#### 10.3.2 Laboratory Variable Changes Relative to Normal Range

Changes relative to normal ranges are presented with shift tables with total number of patients, and number and percent of patients who experienced a shift by treatment group and period. The following categories for shift tables are defined:

• Low: Values which are below the lower reference range limit;

• Normal: Values which are within the lower and upper reference range;

• High: Values which are above the upper reference range limit.

• Absent: No value for measured variable (for urinalysis only)

• Present: Any value obtained for measured variable (for urinalysis only)

For all hematology and clinical chemistry variables, shift tables will be prepared to compare baseline values to the worst in-treatment value. More specifically, for hematology and clinical chemistry, tables presenting the changes from *Low* or *Normal* to *High* and from *High* or *Normal* to *Low* will be provided. For urinalysis variables, shift tables will summarize the number (%) of patients who had "absent" values at baseline and "present" values during the treatment period.

TLF Table: Incidence of hematology laboratory variable changes relative to normal range – Safety Analysis Set

TLF Table: Incidence of chemistry laboratory variable changes relative to normal range – Safety Analysis Set

TLF Table: Incidence of urinalysis variable changes relative to normal range – Safety Analysis Set

## 10.3.3 Data Listings

Data listings will be prepared by treatment group and center for all patients with any abnormal laboratory value at any time-point (including screening, baseline).

TLF Listing: Patients with abnormal laboratory measurements


## 10.3.4 Urinalysis

Incidence of changes in urinalysis will be summarized by treatment. A summary table with number of patients with change from *Absent* at baseline to *Present* during trial will be summarized.

## TLF Table: Incidence of changes from baseline in urinalysis measurements during the trial – Safety Analysis Set

## 10.4 Vital Signs

## 10.4.1 Vital Signs

Baseline for all vital signs analyses will be the values obtained at the last assessment prior to the first dose of IMP. Treatment-emergent vital signs data will include tests completed after the first dose of IMP through the time of residual drug effect. End of trial will include the last post-baseline observation during the trial.

## 10.4.1.1 Summary Statistics

Mean change and mean percentage (%) change from baseline at end of trial will be presented for each vital signs variable. In addition, descriptive statistics, i.e., the number of patients with data, mean (standard deviation), median, minimum, and maximum values, will be presented for observed values and change from baseline at each time-point for each vital signs variable.

TLF Table: Summary of vital signs parameters by visit – Safety Analysis Set

#### 10.4.1.2 Markedly Abnormal Changes

Summary tables will be prepared displaying the number and percentage of patients with normal baseline values who had one or more pre-specified markedly abnormal treatment-emergent value, as defined in Appendix 1.

TLF Table: Incidence of Markedly abnormal vital signs measurements – Safety Analysis Set

#### 10.4.1.3 Data Listings

Data listings will be prepared by center for all patients with any abnormal vital signs value at any time-point (including screening, baseline).

TLF Listing: Patients with Markedly abnormal vital signs measurements

Degarelix, FE 200486 Trial Code: 000108 Statistical Analysis Plan Date: 24 Feb 2021 E-Statistical Analysis Plan-19595; Ver.7.0 Supersedes: 6.0


## 11 Interim Analysis

As the trial was terminated early due to feasibility reasons, planned interims analyses have been cancelled.


## 12 Deviations from Protocol Analysis

List of key secondary endpoints has been revised and testing procedure changed from Holm's to fixed-sequence.

Due to the trial being terminated early due to feasibility reasons, the statistical analysis plan has been reduced. See change log for details.


## 13 References

ADDPLAN, Inc., an Aptiv Solutions Company (2011). ADDPLAN BASE version 6.0 User Manual, Rev. 2. Aptiv Solutions, Cologne, Germany.

Lin, D.Y., Wei, L.J., and Ying, Z. (1993). Checking the Cox model with cumulative sums of martingale-based residuals. *Biometrika* **80**, 557–572.

Prentice RL, Williams BJ and Peterson AV. On the regression analysis of multivariate failure time data. Biometrika 1981;68:373-79.

Wassmer G. Planning and Analyzing Adaptive Group Sequential Survival trials. Biom. J 2006 Aug;48(4):714-29.

Zhao et al., A Multiple Imputation Method for Sensitivity Analyses of Time-To-Event Data With Possibly Informative Censoring. J Biopharm Stat 2014 24(2) 229-253.

Andersen P.K. and Gill, R.D. Cox's Regression Model for Counting Processes: A Large Sample Study. The Annals of Statistics 1982; 4: 1100-1120.

Jennison, C. and Turnbull, B.W. (2000), Group Sequential Methods with Applications to Clinical Trials, New York: Chapman & Hall.

Wei, L.J., Lin, D.Y. and Weissfeld, L. Regression Analysis of Multivariate Incomplete Failure Time Data by Modeling Marginal Distributions. JASA 1989; 408:1065-1073.

Wu, L. and Cook, R.J. Misspecification of Cox regression models with composite endpoints. Stats In Med 2012; 31: 3545-3562.

Blanche, P., Dartigues, J.F. and Jacqmin-Gadda, H. Review and comparison of ROC curve estimators for a time-dependent outcome with marker-dependent censoring. Biometrical J., 55(2013) 5, 687-704.

Hung, H. and Chiang, C. Optimal composite markers for time-dependent receiver operator characteristic curves with censored survival data. Scandinavian Journal of Statistics (2010)37, 664-679.

Uno, H. Cai, T., Tian, L. and Wei, L. Evaluating prediction rules for t-year survivors with censored regression models. JAMA (2007)102, 527-537.

Kalbfleisch, J.D. and Prentice, R.L.(2002) The Statistical Analysis of Failure Time Data, 2<sup>nd</sup> Edition, New York: Wiley.

Therneau, T.M. and Grambsch, P.M. (2000) Modeling Survival Data: Extending the Cox Model, New York: Springer-Verlag.

Degarelix, FE 200486 Trial Code: 000108 Statistical Analysis Plan Date: 24 Feb 2021 E-Statistical Analysis Plan-19595; Ver.7.0 Supersedes: 6.0


## 14 Tables, Listings and Figures

An overview of the tables, listings and figures (TLFs) to be produced is provided in a separate document.


# Appendix 1 Markedly Abnormal Vital Signs and Electrocardiograms (ECGs)

Table 2 Markedly abnormal Criteria for Vital Signs\*

| Variable | Criterion Value | Change from Baseline |
|---|---|---|
| Systolic blood pressure | $\geq 180 \text{ mmHg}$<br>$\leq 90 \text{ mmHg}$ | Increase of≥20 mmHg<br>Decrease of≥20 mmHg |
| Dia stolic blood pressure | ≥ 105 mmHg<br>≤ 50 mmHg | Increase of≥15 mmHg<br>Decrease of≥15 mmHg |
| Pulse rate | ≥ 120 bpm<br>≤ 50 bpm | Increase of≥15 bpm Decrease of≥15 bpm |
| Body weight | None | Increase of≥7% Decrease of≥7% |
| Body temperature | ≥38.3°C | Increase to ≥39.4°C |

<sup>\*</sup> To be identified as markedly abnormal, a treatment value must meet the criterion value and also the specified change from baseline.

Table 3 Abnormal Criteria for Quantitative ECG Data

| Variable | Baseline | Abnormal Treatment-Emergent Value |
|---|---|---|
| ECG heart rate | Normal | ≤ 50 bpm and decrease from baseline of ≥ 15 bpm<br>≥ 120 bpm and increase from baseline of ≥ 15 bpm |
| Duration of PR interval | Normal | ≥ 220 msec |
| Duration of QRS interval | Normal | ≥ 120 msec |
| Duration of QTc interval | Normal | ≥ 450 msec |
| Duration of QTc interval | Normal | ≥ 480 msec |
| Duration of QTc interval | Normal | ≥ 500 msec |
| Duration of QTc interval | Not applicable | Increase from baseline of≥30 msec |
| Duration of QTc interval | Not applicable | Increase from baseline of ≥ 60 msec |


## **Appendix 2 SMQs for AE Medical History of Special Interest**

## Table 4 Cardiovascular Events

| SMQ | SMQ code |
|---------------------------------------------------------|----------|
| Myocardial infarction | 20000047 |
| Ischaemic central nervous system vascular conditions | 20000063 |
| Haemorrhagic central nervous system vascular conditions | 20000064 |
| Embolic and thrombotic events, arterial | 20000082 |
| Other ischaemic heart disease | 20000168 |

## **Table 5** Diabetes Events

| SMQ | SMQ code |
|--------------------------------------------|----------|
| Hyperglycaemia/new onset diabetes mellitus | 20000041 |


## **Appendix 3** ATC codes and MedDRA terms for disease progression

A list of ATC codes for antiandrogens and additional therapies classified as disease progression are defined below. Please note that the list may be non-extensive.

Table 6 ATC Codes for Antiandrogens

| Level 5 codes |
|---------------------|
| L02BB01 Flutamide |
| L02BB02Nilutamide |
| L02BB03Bicalutamide |
| L02BB04Enzalutamide |
| G03HA01 Cyproterone |

Table 7 ATC codes for Additional Therapy

| Level 5 codes |
|---------------------------------|
| L01DB07Mitoxantrone |
| L01CD02Docetaxel |
| L01XX11 Estramustine |
| L01CD01 Paclitaxel |
| L02AA01 Diethylstilbestrol |
| L02AA02 Polyestradiol phosphate |
| L02AA03 Ethinylestradiol |
| L02AA04 Fosfestrol |
| L02AB01 Megestrol |
| L02BG01 Aminoglutethimide |
| L02BX03 Abiraterone |
| G01AF11 Ketoconazole |

Investigators recording of disease progression are marked as a tick-box on the Adverse Event form in the eCRF. The MedDRA terms to be used for radiation and second line treatment are defined below.


Table 8 MedDRA Codes (preferred terms) for Radiation

| 10006089 | Brachytherapy to prostate | PT |
|----------|----------------------------------------|----|
| 10014442 | Electron radiation therapy to prostate | PT |
| 10017683 | Gamma radiation therapy to prostate | PT |
| 10034955 | Photon radiation therapy to prostate | PT |
| 10061544 | Radiotherapy to prostate | PT |
| 10048205 | X-ray therapy to prostate | PT |
| 10014435 | Electron radiation therapy to bone | PT |
| 10017675 | Gamma radiation therapy to bone | PT |
| 10034947 | Photon radiation therapy to bone | PT |
| 10062089 | Radiotherapy to bone | PT |
| 10048197 | X-ray therapy to bone | PT |

 Table 9
 MedDRA Codes (preferred terms) for Second Line Treatment

| 10061916 | Prostatectomy | PT |
|----------|-----------------------------|----|
| 10050756 | Radical prostatectomy | PT |
| 10038961 | Retro-pubic prostatectomy | PT |
| 10042594 | Supra pubic prostatectomy | PT |
| 10044445 | Transurethral prostatectomy | PT |

The following terms are also to be classified as investigators recording of disease progression, in case the investigator did not check the tick-box, but only recorded the AE.

Table 10 MedDRA Codes (preferred terms) for additional classification of investigators recording of disease progression

| 10010264 | Condition a ggravated | PT |
|----------|--------------------------------|----|
| 10061818 | Disea se progression | PT |
| 10061819 | Disea se recurrence | PT |
| 10048669 | Terminal state | PT |
| 10051398 | Malignant neoplasm progression | PT |
| 10027452 | Meta stases to bone | PT |
| 10027459 | Meta stases to lymph nodes | PT |
| 10027457 | Meta stases to liver | PT |
| 10027458 | Meta stases to lung | PT |
| 10027463 | Meta stases to pleura | PT |
| 10062194 | Metastasis | PT |


## **Appendix 4 ATC codes and MedDRA terms for Prohibited Therapy**

A list of ATC codes for prohibited concomitant medication are defined below. Please note that the list may be non-extensive.

Table 11 ATC codes for prohibited concomitant medication

| Level 5 codes |
|---------------------------------|
| L02AB01 Megestrol a cetate |
| G01AF11 Ketoconazole |
| L02BX03 Abiraterone |
| L02BB04Enzalutamide |
| L02BB01Flutamide |
| L02BB02Nilutamide |
| L02BB03Bicalutamide |
| G03HA01 Cyproterone |
| L02AA01 Diethylstilbestrol |
| L02AA02 Polyestradiol phosphate |
| L02AA03 Ethinylestradiol |
| L02AA04 Fosfestrol |

Additionally all substances in the ATC G03 therapeutic subgroup are considered as prohibited concomitant medications.

Table 12 MedDRA code (preffered term) for prohibited therapy

| 10049628 Bilateral orchidectomy | PT |
|---------------------------------|----|
|---------------------------------|----|


## **Appendix 5** Cardiovascular Endpoint Definitions

## **Endpoints / Event definitions**

The cardiovascular endpoint definitions given below are based on the 2014 Definitions for Cardiovascular Endpoint Events in Clinical Trials<sup>1</sup>.

#### 1.1 Death

All deaths will be categorized as Cardiovascular, non-Cardiovascular or Undetermined.

Cardiovascular Death: Cardiovascular Death is defined as death resulting from an acute myocardial infarction, sudden cardiac death, death due to heart failure, death due to stroke, death due to cardiovascular procedures, death due to cardiovascular hemorrhage, and death due to other cardiovascular causes.

**Non-cardiovascular Death:** Non-cardiovascular death is defined as any death that is not thought to be due to a cardiovascular cause (e.g. cancer related death). Non-cardiovascular deaths will also be sub-classified as related to prostate cancer progression or to other causes.

Undetermined Cause of Death: Undetermined cause of death refers to a death not attributable to one of the above categories of cardiovascular death or to a non-cardiovascular cause, due to absence of any information (e.g., the only available information is "patient died"). Undetermined death will be presumed and analyzed as non-cardiovascular deaths on the secondary analysis.

## 1.2 Myocardial Infarction

The adjudication of myocardial infarction as a clinical endpoint will consider the occurrence relative to a percutaneous coronary intervention (PCI) or coronary artery by-pass grafting (CABG). (It will also be consistent with the revised American College of Cardiology (ACC) / European Society of Cardiology (ESC) myocardial infarction definition document.)

In the absence of a PCI or CABG, a spontaneous myocardial infarction is defined as:



For patients having a PCI, a myocardial infarction will be defined as:

CK-MB (or troponin I/T or CK in the absence of CK-MB) >3 x ULN for samples obtained within 24 hours of the procedure if the baseline values were normal or at least a 50% increase

over elevated baseline values that were stable or decreasing or development of new pathological Q waves (>0.04 seconds) in at least 2 contiguous leads in the absence of LBBB on the ECG. Symptoms of cardiac ischemia are not required.

After CABG surgery, a myocardial infarction is defined as either:

CK-MB (or CK in the absence of CK-MB) >5 x ULN for samples obtained within 24 hours of the procedure with development of new pathological Q waves in at least 2 contiguous leads in the absence of LBBB on the ECG.

CK-MB (or CK in the absence of CK-MB) > 10 x ULN for samples obtained within 24 hours of the procedure with or without development of new pathological Q waves in at least 2 contiguous leads in the absence of LBBB on the ECG.

Note: For institutions that report an 'intermediate' or 'equivocal' range for biomarker elevation that is not definitively associated with myocardial necrosis or infarction then the ULN should be the lower value for the necrosis or infarct range, not the 'equivocal' or 'intermediate' range lower value.

## 1.3 Unstable Angina Requiring Hospitalization

## 1.4 Cerebrovascular Accident (Stroke)

Stroke is defined as an acute focal neurological deficit of sudden onset that is not due to an identifiable non-vascular cause (i.e. brain tumor, trauma, brain procedures, metabolic condition)

Degarelix, FE 200486 Trial Code: 000108 Statistical Analysis Plan Date: 24 Feb 2021 E-Statistical Analysis Plan-19595; Ver.7.0 Supersedes: 6.0


a) that is not reversible within 24 hours or results in death (in <24 hours)

or

b) that resolves in <24 hours and is accompanied by clear evidence of a new stroke on cerebral brain imaging studies (brain Computed tomography [CT] or Magnetic Resonance Imaging [MRI] scans)

#### Classification:

**Ischemic Stroke:** is defined as an acute episode of focal cerebral, spinal, or retinal dysfunction caused by central nervous system (CNS) infarction.

Note: Hemorrhage may be a consequence of ischemic stroke. In this situation, the stroke is an ischemic stroke with hemorrhagic transformation and not a hemorrhagic stroke.

**Hemorrhagic Stroke:** is defined as an acute episode of focal or global cerebral or spinal dysfunction caused by intraparenchymal, intraventricular, or subarachnoid hemorrhage.

Note: Subdural hematomas without new neurologic symptoms are intracranial hemorrhagic events and not strokes.

**Undetermined Etiology:** is defined as an acute episode of focal or global neurological dysfunction caused by presumed brain, spinal cord, or retinal vascular injury as a result of hemorrhage or infarction but with insufficient information to allow categorization as either ischemic or hemorrhagic.

Hicks KA, Tcheng JE, Bozkurt B, Chaitman BR, Cutlip DE, Farb A, et al. 2014 ACC/AHA Key Data Elements and Definitions for Cardiovascular Endpoint Events in Clinical Trials: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Data Standards (Writing Committee to Develop Cardiovascular Endpoints Data Standards). J Am Coll Cardiol 2015 Jul 28;66(4):403-69.